CLINICAL TRIAL: NCT02164305
Title: The Effects of Exercise Training on Shoulder Neuromuscular Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07252013.032
Record Dates: First submitted 2014-05-21; First posted 2014-06-16 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Shoulder Impingement
Keywords: Rotator cuff muscle; Excitability; Proprioception; Kinematics; Muscle activity; Electromyography
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Strengthening group (Experimental): 4-week exercise training, 3 times a week, 30 minutes per visit.
  Interventions: Other: Strengthening group
- Neuromuscular group (Experimental): 4-week exercise training, 3 times a week, 30 minutes per visit
  Interventions: Other: Neuromuscular group
- Control (Sham Comparator): Only have 2 assessments.
  Interventions: Other: Control

INTERVENTIONS:
Other: Strengthening group — Open-chain exercise for rotator cuff and scapular muscles
  Arms: Strengthening group
Other: Neuromuscular group — Closed-chain exercise for shoulder muscles
  Arms: Neuromuscular group
Other: Control — No exercise training
  Arms: Control

SUMMARY:
Dynamic control of the rotator cuff muscles plays an important role in stabilizing the shoulder during motion. Impairment in the neuromuscular control of these muscles may to lead to injury and pain. Rehabilitation programs have moderate success in decreasing pain and improving shoulder function. While most of these programs target the rotator cuff, it is still unknown if they serve to improve the neuromuscular control of the rotator cuff muscles. The rehabilitation may induce neurological and physiologic changes in neuromuscular structures and thus alter the neuromuscular control of the entire shoulder complex. Kinematics and electromyographic (EMG) activities have been widely used to study neuromuscular control. However, corticospinal excitability, which has been widely examined in the patients with neurological disorders, provides a more detailed account of central control from the primary motor cortex through the spinal cord to the muscles. This assessment of neuromuscular control will serve to illuminate the ability of the shoulder muscles to handle the stress from activities such as overhead sports activities and carrying or lifting heavy objects. This approach could be used to help design efficient training program for athletes and effective rehabilitation program for patients with shoulder injuries. The purpose of the proposed study is to investigate the effect of exercise treatment effect on the proprioception, kinematics, EMG and corticospinal excitability of shoulder muscles, including the deltoid and rotator cuff muscles.

DETAILED DESCRIPTION:
Significance

The human shoulder complex sacrifices stability in exchange for a large range of motion necessary for hand manipulation. Due to the inherent instability of the bony congruence and ligament constraint, dynamic control of the muscles plays an important role in stabilizing the shoulder during motion. The rotator cuff muscles serve as the chief stabilizer of the shoulder joint, while the deltoid provides most of the torque necessary for motion. Therefore, the coordination of the deltoid and the rotator cuff muscles is essential for smooth and efficient shoulder function. Impairment in the neuromuscular control of these muscles may to lead to injury and pain. Consequently, rehabilitation programs aim to restore the normal neuromuscular control of these shoulder muscles in order to help decrease pain and improve shoulder function. Although rehabilitation programs have demonstrated positive effects on pain decrease and functional improvement, it is still unknown if they serve to improve the neuromuscular control of the shoulder muscles.

While the deltoid provides most of the torque necessary to elevation the shoulder, it can also produce a superiorly directly force on the glenoid. This shear force tends to pull the humeral head superiorly, which can result in a decrease in the subacromial space. When the rotator cuff muscles function properly, the line of action of the rotator cuff muscles result in a centering force, which can help maintain the humeral head in the center of the glenoid fossa. However, it has been hypothesized that if the rotator cuff muscles are not able to produce sufficient force during arm movement, the superior shear force produced by the deltoid results in humeral head superior translation. This abnormal displacement can result in impingement of subacromial tissues and ultimately leading to tissue injury and pain.

Traditionally, shoulder rehabilitation programs focus on strengthening the rotator cuff muscles by using shoulder movement in which the rotator cuff muscles show high muscle activity. However, although these activities lead to a strengthening of the rotator cuff, what is unknown is whether the repetitive stress imposed on the rotator cuff results in neuromuscular adaptations that will help counteract the deltoid shear force.

This stress of rehabilitation may induce the neurological and physiologic changes in neuromuscular structures and thus alters the neuromuscular control of the entire shoulder complex. Kinematics and electromyographic (EMG) measurements have been widely used to study neuromuscular control. While kinematic measures show movement patterns, EMG demonstrates the timing, sequence, and magnitude of the muscle firing. Abnormal kinematics and EMG patterns have been demonstrated in patients with shoulder impingement. Measuring parameters of neuromuscular control can lead to a better understanding of the underlying mechanism of shoulder exercise training and how the neuromuscular structures adapt to the stress of the exercise training. More specifically, these assessments can be used to assess whether a rehabilitation program results in a positive adaptation that can help the shoulder muscles handle the stress from activities such as overhead sports activities and carrying or lifting heavy objects. Ultimately, this could be used to design more efficient training program for athletes and effective rehabilitation program for patients with shoulder injuries.

Innovation

When shoulder neuromuscular control is investigated in the fields of biomechanics, orthopaedic rehabilitation, and sports, the focus is generally on kinematics and EMG. These kinematics and EMG parameters represent how the shoulder complex is controlled during movement as the result of motor command execution. Corticospinal excitability, which has been widely examined in patients with neurological disorders, has also been recently applied in biomechanics, orthopaedic rehabilitation, and sports fields. Corticospinal excitability represents the efficacy of neural transmission along the corticospinal pathway. In addition to neurological impairment, orthopaedic injury and pain can also affect corticospinal excitability. For example, in subjects with non-traumatic shoulder instability, the lower trapezius demonstrates decreased excitability. Also, experimental tonic muscle pain over the first dorsal interosseous results in inhibition of cortical and spinal excitability. Similarly, experimentally-induced acute low lumbar pain is associated with different effects on trunk muscles. The deep abdominal muscles, such as the transversus abdominis, showed reduced corticospinal excitability. In contract, more superficial muscles, such as the lumbar erector spinae and external oblique abdominis, demonstrated increased excitability. In addition to kinematics and EMG measurements, which demonstrate the overall motor strategy, the corticospinal excitability is another promising parameter to investigate the details about how the deltoid and rotator cuff muscles are controlled from the primary motor cortex through the spinal cord to the muscle.

While consistent evidence suggests that motor skill training is associated with increased excitability, the effects of strength training on corticospinal excitability are still not well known and may depend on the muscles and training task. The training of neuromuscular control may be associated with both motor learning and strength training. The control and firing pattern may be directly re-learned consciously, which involves increases in strength and motor learning. Since it is associated with a learning process, excitability may increase after training. It has been shown that changes in the excitability are correlated with a motor learning effect, so that changes in excitability after training may be correlated with changes of rotator cuff EMG. After repetitive practice, the conscious movement patterns may become automatic thus changing the EMG pattern of rotator cuff activation.

The purposes of the study are to (1) investigate the effect of exercise training on the neuromuscular control of shoulder complex in healthy subjects, including kinematics, EMG and corticospinal excitability, and (2) to examine the relationship between the corticospinal excitability, EMG and force measures. The results of the study may help to understand the underlying neurological and biomechanic mechanism of exercise training and help to design the training or rehabilitation protocols for the athletes or the patient with shoulder injuries.

Approach

A randomized controlled experimental design will be used to investigate the effect of rotator cuff exercise. Healthy subjects will be recruited and randomly assigned to two groups, exercise and control groups.

All measures will be made twice, before and after a four-week treatment. Fine-wire electromyography (EMG) electrodes will be inserted into the supraspinatus and infraspinatus muscles of the rotator cuff. Surface EMG electrodes will be used for the middle deltoid and scapular muscles. Transcranial magnetic stimulation (TMS) will be used to assess the corticospinal excitability of the deltoid and rotator cuff muscles. A flat double-coil stimulation coil will be used to provide a single-pulse stimulus over the motor cortex, approximately 4 cm lateral of the bisection of the mid line and the biauricular line. Electromagnetic tracking sensors will be attached to the arm, scapula and thorax to measure shoulder kinematics.

The parameters of corticospinal excitability will also measured when the arm is at 90° of elevation with a baseline muscle contraction level of 10% maximum voluntary contraction (MVC). TMS stimulation intensity will be set at 10% below threshold and increased in 5% increments until the response saturates. Five stimuli will be delivered at each intensity of stimulation. The peak-to-peak amplitude of the motor evoked potential (MEP) will be measured and averaged across the five trials at each intensity. The curve of the relationship between stimulation intensity and the MEP amplitude is sigmoidal and will be fit with the Boltzmann equation.

MEP(s) = MEPmax/(1+ e^(m(S - 50s)))

In this equation, MEP(s) is the amplitude of motor evoked potential, MEPmax is the maximum MEP amplitude, m is the slope of the function, and S50 is the stimulus intensity at which the MEP is 50% of MEPmax. The peak slope of the function occurs at S50. The threshold of the curve is the x-intercept of the tangent to the function at the point of maximal slope.

Three parameters, MEPmax, m, and x-intercept threshold, will be used to model the corticospinal excitability, which provides a more details of the excitability of the corticospinal tract. The value of x-intercept threshold is similar to the motor threshold and represents the stimulus intensity needed to activate the most excitable corticospinal elements and motoneurons. The slope indicates the recruitment efficiency (gain) of the corticospinal tract. The MEPmax reflects the balance between excitatory and inhibitory components of the corticospinal tract.

Scapular and humeral kinematics and the dynamic EMG of rotator cuff and deltoid muscles will be recorded during three trials of arm elevation at scapular plane. The root mean square EMG data will be calculated over four 30° increments of motion during arm elevation from 0° to 120°. Scapular kinematics will be presented at 30°, 60°, 90° and 120° of humeral elevation.

The subjects will be tested the shoulder proprioception. They will wear a goggle, which will give the visual cues to guide them to reach the target. Three target positions will be presented: humerothoracic elevation angles of 50°, 70°, and 90° in the scapular plane. The subjects will be instructed to reach the target again without any visual cues after relaxing their arms at the side. The errors between the target angle and the angle they returned will be calculated.

Both treatment programs will last four weeks. The subjects in the exercise group will have standard rehabilitation exercise for the shoulder impingement syndrome. The exercise will be based on a previous treatment study conducted by Dr. Karduna and will be modified to emphasize on facilitation and strengthening the rotator cuff muscles. The subjects in the control group will receive no exercise. The control subjects will be asked to maintain their regular activities and only have two assessments.

A two-way mixed-design analysis of variance (ANOVA) will be used to examine the differences in neuromuscular control following the treatment between the control and exercise groups. The dependent variables will be the changes of kinematics, EMG and excitability following the treatment. The independent variables will be humeral elevation angles and groups. The correlation between changes of TMS measures, the EMG measures, and the forces will be examined by with a correlation analysis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects

Exclusion Criteria:

* Less than 135 degrees of active humeral elevation in the scapular plane
* Prior shoulder and cervical surgery
* Presence of shoulder and neck pain
* Had history of head, cervical or shoulder pain or pathology
* Stroke and neurological impairment
* History of seizures
* Taking anti-seizure and anti-depressive medication
* With pacemaker and other magnetic implant
* Pregnancy
* Athletes performing upper extremity exercise

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2014-05; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in muscle activity of rotator cuff and scapular muscles at 4 weeks | Baseline and 4 weeks

SECONDARY OUTCOMES:
Change from baseline in elevation force at 4 weeks | Baseline and 4 weeks
Change from baseline in proprioception errors at 4 weeks | Baseline and 4 weeks
Change from baseline in the amplitude of motor evoked potential of rotator cuff at 4 weeks | Baseline and 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Karduna, PhD, Study Director — Department of Human Physiology at University of Oregon
Locations (1):
- University of Oregon, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No